CLINICAL TRIAL: NCT00549549
Title: A Phase 3, Randomized, Double-Blind, Multicenter, Active-Controlled Trial To Evaluate The Efficacy And Safety Of Celecoxib (Celebrex®) And Indomethacin In The Treatment Of Moderate To Severe Acute Gouty Arthritis
Brief Title: Celebrex In Acute Gouty Arthritis Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3191219
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Arthritis, Gouty
MeSH Terms: conditions — Arthritis, Gouty | interventions — Indomethacin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Indomethacin
- 2 (Experimental)
  Interventions: Drug: Celecoxib
- 3 (Experimental)
  Interventions: Drug: Celecoxib
- 4 (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Indomethacin — indomethacin 50 mg three times a day (TID) for 8 days.
  Arms: 1
Drug: Celecoxib — An initial dose of celecoxib 800 mg followed by a second dose of 400 mg 12 hours later on Day 1 (celecoxib 800/400 mg regimen) and continuing 400 mg two times a day (BID) for 7 days.
  Arms: 2
Drug: Celecoxib — An initial dose of celecoxib 400 mg followed by a second dose of 200 mg 12 hours later (celecoxib 400/200 mg regimen) and continuing 200 mg two times a day (BID) for 7 days.
  Arms: 3
Drug: Celecoxib — Celecoxib 50 mg two times a day (BID) for 8 days
  Arms: 4

SUMMARY:
This is a multicenter, double-blind, double-dummy, randomized, active-controlled study that will include an 8-day treatment period followed by a 1-week follow-up period in patients experiencing symptoms of an acute exacerbation of gouty arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Acute gouty arthritis meeting the American College of Rheumatology (ACR) criteria for acute arthritis of primary gout;
* Onset of pain from an acute gouty arthritis attack within 48 hours prior to Screening/Baseline (Visit 1);
* A rating of moderate, severe, or extreme (2, 3, or 4, respectively) on the Patient's assessment of pain intensity in the index joint (5-point scale:0-4) at Screening/Baseline.

Exclusion Criteria:

* Diagnosis of any other type of arthritis including those types suspected of being infectious in origin in the index joint or presence of any acute trauma of the index joint. Patients with osteoarthritis will be included as long as it is mild or moderate (according to investigator's criteria) and it does not affect the index joint;
* Acute polyarticular gout involving greater than 4 joints or chronic gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (40):
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Luis Obispo, California
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Northglenn, Colorado
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Dunwoody, Georgia
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Columbus, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Willoughby Hills, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Havertown, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Canada (9):
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Colombia (2):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bucaramanga, Santander Department
- Costa Rica (2):
  - Pfizer Investigational Site, Cartago
  - Pfizer Investigational Site, Heredia
- Mexico (3):
  - Pfizer Investigational Site, México, D.F.
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Pfizer Investigational Site, Lima, Peru
- Philippines (4):
  - Pfizer Investigational Site, Lipa City, Batangas
  - Pfizer Investigational Site, Las Piñas
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Petrozavodsk
  - Pfizer Investigational Site, Saint Petersburg
- South Korea (2):
  - Pfizer Investigational Site, Suwon, Kyeongki-do
  - Pfizer Investigational Site, Daegu
- Pfizer Investigational Site, Seville, Spain
- Taiwan (3):
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Phayathai, Bangkok
  - Pfizer Investigational Site, Khon Kaen

REFERENCES:
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191219&StudyName=Celebrex%20In%20Acute%20Gouty%20Arthritis%20Study

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 443 participants were screened, of which 402 participants were assigned to treatment and 400 received treatment. One participant (indomethacin 50 mg) was not treated as they were no longer willing to participate in the study, and one participant (celecoxib 800/400 mg) was not treated due to due to insufficient drug quantity at site.
Groups:
- Celecoxib 50 mg: Participants received Celecoxib 50 mg twice daily for 8 days
- Celecoxib 400/200 mg: An initial dose of celecoxib 400 mg followed by a second dose of 200 mg 12 hours later on Day 1 (celecoxib 400/200 mg regimen) and continuing 200 mg twice daily for 7 days.
- Celecoxib 800/400 mg: An initial dose of celecoxib 800 mg followed by a second dose of 400 mg 12 hours later on Day 1 (celecoxib 800/400 mg regimen) and continuing 400 mg twice daily for 7 days.
- Indomethacin 50 mg: Indomethacin 50 mg three times daily for 8 days.
Period: Overall Study
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Started | 101 | 99 | 99 | 103
Treated | 101 | 99 | 98 | 102
Completed | 77 | 77 | 82 | 78
Not Completed | 24 | 22 | 17 | 25
Not completed — Adverse Event | 5 | 3 | 1 | 9
Not completed — Lack of Efficacy | 9 | 6 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 0
Not completed — Other | 9 | 9 | 9 | 11
Not completed — Randomized but not treated | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg | Total
Number analyzed (Participants) | 101 | 99 | 98 | 102 | 400
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 84 | 83 | 86 | 88 | 341
  >=65 years | 17 | 16 | 12 | 14 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 8 | 7 | 34
  Male | 91 | 90 | 90 | 95 | 366
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 53 | 64 | 54 | 55 | 226
  Black | 11 | 3 | 10 | 9 | 33
  Asian | 22 | 18 | 19 | 19 | 78
  Other | 15 | 14 | 15 | 19 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 2 in Patient's Assessment of Pain Intensity
Description: The Patient's Pain Intensity in the Index Joint for the prior 24 hours was assessed by completion of the following 5 point scale: My pain over the past 24 hours has been: None (0), Mild (1), Moderate (2), Severe (3), or Extreme (4).
Time Frame: Baseline and Day 2
Population: Intent to treat (ITT): defined to be all subjects who were randomized, took at least 1 dose of study medication and had at least one post baseline evaluation; and Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 3.03 (0.67) | 2.73 (0.62) | 2.84 (0.69) | 2.83 (0.76)
  Change at Day 2 | -1.14 (1.10) | -1.23 (0.97) | -1.51 (1.11) | -1.62 (0.97)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; This was the primary analysis. The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular) and treatment group and region as factors, and the Patient's Assessment of Pain Intensity (for the prior 24 hours) at Baseline as a covariate; Test type: Superiority or Other; ANCOVA; Median Difference (Final Values) = -0.46, 95% CI 2-sided [-0.74 to -0.18], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Test type: Superiority or Other; ANCOVA; Median Difference (Final Values) = -0.24, 95% CI 2-sided [-0.52 to 0.04], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [0.29 to 0.84], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.05 to 0.60], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.17 to 0.39], Standard Error of Mean 0.14

2. Secondary Outcome: Change From Baseline in Physician's Assessment of the Index Joint on Days 5, 9, and 14/Early Termination: Tenderness
Description: Tenderness was assessed on the basis of palpation or passive motion using a 4 point scale with the following ratings: the patient had no tenderness (0), the patient complained of pain (1), the patient complained of pain and winced (2) and the patient complained of pain, winced, and withdrew (3).
Time Frame: Baseline, Day 5, Day 9, and Day 14/Early Termination
Population: Intent to treat (defined to be all subjects who were randomized, took at least 1 dose of study medication and had at least one post baseline evaluation, ITT) and LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 2.39 (0.72) | 2.15 (0.75) | 2.26 (0.65) | 2.13 (0.70)
  Change at Day 5 | -1.44 (0.96) | -1.39 (0.89) | -1.58 (0.93) | -1.52 (0.86)
  Change at Day 9 | -1.75 (0.98) | -1.64 (0.93) | -1.84 (0.92) | -1.65 (0.87)
  Change at Day 14/Early Termination | -1.74 (1.09) | -1.66 (1.01) | -1.94 (0.88) | -1.64 (0.93)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 5 analysis. The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular) and treatment group as factors, and the Patient's Assessment of Pain Intensity (for the prior 24 hours) at Baseline as a covariate; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.29 to 0.14], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.42 to 0.02], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.04 to 0.47], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.04 to 0.39], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.16 to 0.27], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.26 to 0.16], Standard Error of Mean 0.11
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.40 to 0.03], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.11 to 0.32], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.16 to 0.27], Standard Error of Mean 0.11
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.30 to 0.13], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.33 to 0.10], Standard Error of Mean 0.11
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.53 to -0.11], Standard Error of Mean 0.11
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day /early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.05 to 0.37], Standard Error of Mean 0.11
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.17 to 0.25], Standard Error of Mean 0.11
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.38 to 0.05], Standard Error of Mean 0.11

3. Secondary Outcome: Change From Baseline in Physician's Assessment of the Index Joint on Days 5, 9, and 14/Early Termination: Swelling
Description: Swelling was assessed using a 4 point scale with the following ratings: none (0), palpable (1), visible (2), and bulging beyond joint margins (3)
Time Frame: Baseline, Days 5, 9 and 14/Early Termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 2.16 (0.73) | 2.08 (0.65) | 2.09 (0.65) | 2.01 (0.75)
  Change at Day 5 | -1.22 (1.09) | -1.21 (1.05) | -1.27 (0.97) | -1.20 (0.96)
  Change at Day 9 | -1.47 (1.18) | -1.54 (1.00) | -1.62 (0.95) | -1.58 (0.94)
  Change at Day 14/Early Termination | -1.55 (1.18) | -1.63 (0.98) | -1.78 (0.97) | -1.58 (0.94)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.29 to 0.22], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.35 to 0.16], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.17 to 0.34], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.20 to 0.30], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 5 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.26 to 0.25], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.36 to 0.11], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.44 to 0.04], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.01 to 0.46], Standard Error of Mean 0.12
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.14 to 0.33], Standard Error of Mean 0.12
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 9 analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.22 to 0.26], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.38 to 0.10], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.52 to -0.04], Standard Error of Mean 0.12
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.08 to 0.39], Standard Error of Mean 0.12
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.22 to 0.26], Standard Error of Mean 0.12
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 14/early termination analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.36 to 0.12], Standard Error of Mean 0.12

4. Secondary Outcome: Number of Participants With Redness Present According to Physician's Assessment of the Index Joint on Day 5, Day 9, and Day 14/Early Termination
Description: Redness was assessed by the physician as present or absent.
Time Frame: Baseline, Day 5, Day 9 and Day 14/Early Termination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants
  Baseline | 84 | 88 | 79 | 85
  Day 5 | 27 | 29 | 26 | 23
  Day 9 | 12 | 15 | 13 | 11
  Day 14/Early termination | 15 | 15 | 7 | 13
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 5 analyses. Pairwise p-values are presented, calculated using Cochran-Mantel-Haenszel statistics, stratified by number of affected joints [1 or >1]) and region; Test type: Superiority or Other; p = 0.6402, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.9739, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.4581, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.2962, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.4951, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.4957, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.8364, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.6892, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.4110, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.5981, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.9317, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.0831, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.5747, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.6204, Cochran-Mantel-Haenszel
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 14/Early Termination analysis; Test type: Superiority or Other; p = 0.2556, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants With Warmth Present According to Physician's Assessment of the Index Joint on Day 5, Day 9, and Day 14
Description: Warmth was assessed by the physician as present or absent.
Time Frame: Baseline, Day 5, Day 9 and Day 14
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants
  Baseline | 89 | 91 | 91 | 88
  Day 5 | 25 | 16 | 22 | 21
  Day 9 | 13 | 8 | 9 | 11
  DAY 14/E_TERM | 19 | 7 | 11 | 15
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1444, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.7532, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.4722, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.3878, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; p = 0.6717, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.3098, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.4356, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.5703, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.4986, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; p = 0.7855, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.0169, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.1353, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.3690, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.0787, Cochran-Mantel-Haenszel
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 14/Early Termination analyses; Test type: Superiority or Other; p = 0.5687, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Intensity
Description: The Patient's assessment of pain for the prior 24 hours was assessed by completion of the following 5 point scale: My pain over the past 24 hours has been: None (0), Mild (1), Moderate, (2), Severe (3), and Extreme (4).
Time Frame: Baseline, Day 2 to Day 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 3.03 (0.67) | 2.73 (0.62) | 2.84 (0.69) | 2.83 (0.76)
  Change at Day 1 | -0.65 (0.87) | -0.85 (0.86) | -1.06 (1.08) | -1.10 (0.92)
  Change at Day 2 | -1.14 (1.10) | -1.23 (0.97) | -1.51 (1.11) | -1.62 (0.97)
  Change at Day 3 | -1.32 (1.15) | -1.42 (0.98) | -1.78 (1.09) | -1.84 (0.97)
  Change at Day 4 | -1.52 (1.16) | -1.60 (0.98) | -1.96 (1.08) | -2.02 (1.00)
  Change at Day 5 | -1.52 (1.16) | -1.67 (1.04) | -2.05 (1.10) | -2.04 (1.03)
  Change at Day 6 | -1.68 (1.15) | -1.84 (1.05) | -2.12 (1.06) | -2.11 (1.01)
  Change at Day 7 | -1.79 (1.23) | -1.90 (1.16) | -2.29 (1.05) | -2.15 (1.02)
  Change at Day 8 | -1.88 (1.26) | -1.95 (1.12) | -2.30 (0.98) | -2.16 (1.04)
  Change at Day 9 | -1.86 (1.27) | -1.96 (1.12) | -2.24 (1.04) | -2.19 (1.08)
  Change at Day 10 | -1.90 (1.27) | -1.99 (1.13) | -2.23 (1.13) | -2.17 (1.01)
  Change at Day 11 | -1.89 (1.31) | -1.94 (1.13) | -2.22 (1.15) | -2.15 (1.02)
  Change at Day 12 | -1.93 (1.32) | -1.95 (1.18) | -2.27 (1.09) | -2.07 (1.07)
  Change at Day 13/Early termination | -1.91 (1.34) | -1.95 (1.18) | -2.27 (1.08) | -1.98 (1.11)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular), region and treatment group as factors, and the Patient's Assessment of Pain Intensity at Baseline as a covariate; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.60 to -0.10], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 1 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.75 to -0.25], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 1 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [0.29 to 0.78], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 1 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.06 to 0.44], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 1 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.21 to 0.28], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 2 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.52 to 0.04], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 2 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.74 to -0.18], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 2 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [0.29 to 0.84], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 2 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.05 to 0.60], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 2 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.17 to 0.39], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 3 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.53 to 0.03], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 3 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.83 to -0.26], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 3 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.32 to 0.88], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 3 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [0.08 to 0.64], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 3 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.22 to 0.34], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 4 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.56 to -0.00], Standard Error of Mean 0.14
Statistical Analysis 17: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 4 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.84 to -0.28], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 4 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [0.35 to 0.90], Standard Error of Mean 0.14
Statistical Analysis 19: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 4 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [0.07 to 0.62], Standard Error of Mean 0.14
Statistical Analysis 20: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 4 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.21 to 0.34], Standard Error of Mean 0.14
Statistical Analysis 21: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 5 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.64 to -0.07], Standard Error of Mean 0.14
Statistical Analysis 22: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 5 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-0.94 to -0.38], Standard Error of Mean 0.14
Statistical Analysis 23: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.37 to 0.93], Standard Error of Mean 0.14
Statistical Analysis 24: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.02 to 0.57], Standard Error of Mean 0.14
Statistical Analysis 25: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 5 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.29 to 0.27], Standard Error of Mean 0.14
Statistical Analysis 26: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 6 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.65 to -0.10], Standard Error of Mean 0.14
Statistical Analysis 27: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 6 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.84 to -0.29], Standard Error of Mean 0.14
Statistical Analysis 28: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 6 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.29 to 0.83], Standard Error of Mean 0.14
Statistical Analysis 29: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 6 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.08 to 0.46], Standard Error of Mean 0.14
Statistical Analysis 30: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 6 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.28 to 0.26], Standard Error of Mean 0.14
Statistical Analysis 31: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 7 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.61 to -0.04], Standard Error of Mean 0.15
Statistical Analysis 32: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 7 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.92 to -0.34], Standard Error of Mean 0.15
Statistical Analysis 33: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 7 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [0.21 to 0.78], Standard Error of Mean 0.14
Statistical Analysis 34: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 7 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.11 to 0.45], Standard Error of Mean 0.14
Statistical Analysis 35: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 7 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.42 to 0.15], Standard Error of Mean 0.14
Statistical Analysis 36: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 8 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.57 to -0.00], Standard Error of Mean 0.14
Statistical Analysis 37: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 8 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.84 to -0.27], Standard Error of Mean 0.14
Statistical Analysis 38: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 8 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.14 to 0.70], Standard Error of Mean 0.14
Statistical Analysis 39: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 8 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.15 to 0.41], Standard Error of Mean 0.14
Statistical Analysis 40: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 8 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.42 to 0.14], Standard Error of Mean 0.14
Statistical Analysis 41: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 9 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.61 to -0.02], Standard Error of Mean 0.15
Statistical Analysis 42: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 9 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.82 to -0.23], Standard Error of Mean 0.15
Statistical Analysis 43: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.18 to 0.76], Standard Error of Mean 0.15
Statistical Analysis 44: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.13 to 0.44], Standard Error of Mean 0.15
Statistical Analysis 45: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 9 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.35 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 46: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 10 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.59 to 0.01], Standard Error of Mean 0.15
Statistical Analysis 47: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 10 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.76 to -0.16], Standard Error of Mean 0.15
Statistical Analysis 48: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 10 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.10 to 0.69], Standard Error of Mean 0.15
Statistical Analysis 49: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 10 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.18 to 0.41], Standard Error of Mean 0.15
Statistical Analysis 50: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 10 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.36 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 51: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 11 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.56 to 0.05], Standard Error of Mean 0.15
Statistical Analysis 52: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 11 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.77 to -0.17], Standard Error of Mean 0.15
Statistical Analysis 53: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 11 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.10 to 0.69], Standard Error of Mean 0.15
Statistical Analysis 54: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 11 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.16 to 0.44], Standard Error of Mean 0.15
Statistical Analysis 55: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 11 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.37 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 56: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 12 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.53 to 0.09], Standard Error of Mean 0.16
Statistical Analysis 57: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 12 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.77 to -0.15], Standard Error of Mean 0.16
Statistical Analysis 58: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 12 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.04 to 0.57], Standard Error of Mean 0.15
Statistical Analysis 59: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 12 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.25 to 0.36], Standard Error of Mean 0.15
Statistical Analysis 60: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 12 analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.50 to 0.11], Standard Error of Mean 0.16
Statistical Analysis 61: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 13/Early Termination analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.56 to 0.07], Standard Error of Mean 0.16
Statistical Analysis 62: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 13/Early Termination analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.81 to -0.19], Standard Error of Mean 0.16
Statistical Analysis 63: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 13/Early Termination analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.10 to 0.51], Standard Error of Mean 0.16
Statistical Analysis 64: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 13/Early Termination analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.35 to 0.26], Standard Error of Mean 0.16
Statistical Analysis 65: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 13/Early Termination analyses; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.60 to 0.01], Standard Error of Mean 0.16

7. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Intensity on Day 1
Description: The patient's assessment of pain was assessed by completion of the following 5 point scale: my pain at this time is none (0), mild (1), moderate, (2), severe (3), and extreme (4).
Time Frame: Baseline, 2, 4, 8, 12 hours postdose Day 1, Day 2 (24 hours and 32 hours post first dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 3.03 (0.67) | 2.73 (0.62) | 2.84 (0.69) | 2.83 (0.76)
  Change at Day 1, 2 HR | -0.32 (0.75) | -0.28 (0.67) | -0.45 (0.77) | -0.57 (0.88)
  Change at Day 1, 4 HR | -0.53 (0.82) | -0.54 (0.69) | -0.70 (0.90) | -0.81 (0.92)
  Change at Day 1, 8 HR | -0.64 (0.92) | -0.58 (0.73) | -0.87 (1.05) | -0.98 (0.94)
  Change at Day 1, 12 HR | -0.73 (1.02) | -0.75 (0.79) | -1.02 (1.11) | -1.09 (0.96)
  Change at Day 2, 0 HR | -0.93 (1.00) | -0.98 (0.88) | -1.15 (1.14) | -1.26 (0.93)
  Change at Day 2, 8 HR | -1.08 (1.07) | -1.07 (0.96) | -1.31 (1.03) | -1.46 (0.93)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular) and treatment group as factors, and the Patient's Assessment of Pain Intensity at Baseline as a covariate; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.28 to 0.14], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 1, 2 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.39 to 0.03], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 1, 2 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [0.11 to 0.52], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 1, 2 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.04 to 0.45], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 1, 2 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.08 to 0.34], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 1, 4 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.37 to 0.08], Standard Error of Mean 0.11
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 1, 4 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.48 to -0.03], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 1, 4 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [0.14 to 0.58], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 1, 4 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.00 to 0.44], Standard Error of Mean 0.11
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 1, 4 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.11 to 0.34], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 1, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.32 to 0.17], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 1, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.56 to -0.06], Standard Error of Mean 0.13
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 1, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.18 to 0.67], Standard Error of Mean 0.12
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 1, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [0.11 to 0.59], Standard Error of Mean 0.12
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 1, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.13 to 0.36], Standard Error of Mean 0.12
Statistical Analysis 16: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 1, 12 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.42 to 0.10], Standard Error of Mean 0.13
Statistical Analysis 17: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 1, 12 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.63 to -0.11], Standard Error of Mean 0.13
Statistical Analysis 18: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 1, 12 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.19 to 0.70], Standard Error of Mean 0.13
Statistical Analysis 19: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 1, 12 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.03 to 0.55], Standard Error of Mean 0.13
Statistical Analysis 20: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 1, 12 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.18 to 0.34], Standard Error of Mean 0.13
Statistical Analysis 21: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 2, 0 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.46 to 0.07], Standard Error of Mean 0.13
Statistical Analysis 22: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 2, 0 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.57 to -0.04], Standard Error of Mean 0.14
Statistical Analysis 23: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 2, 0 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.16 to 0.68], Standard Error of Mean 0.13
Statistical Analysis 24: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 2, 0 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.04 to 0.49], Standard Error of Mean 0.13
Statistical Analysis 25: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 2, 0 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.15 to 0.38], Standard Error of Mean 0.13
Statistical Analysis 26: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Day 2, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.40 to 0.14], Standard Error of Mean 0.14
Statistical Analysis 27: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Day 2, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.59 to -0.05], Standard Error of Mean 0.14
Statistical Analysis 28: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Day 2, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.20 to 0.74], Standard Error of Mean 0.14
Statistical Analysis 29: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Day 2, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [0.08 to 0.61], Standard Error of Mean 0.13
Statistical Analysis 30: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Day 2, 8 hours postdose; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.11 to 0.42], Standard Error of Mean 0.14

8. Secondary Outcome: Change From Baseline in Time Weighted Average of Patient's Assessment of Pain Intensity Over 8, 12, and 24 Hours
Description: Time weighted average over 8 (TWA-8), 12 (TWA-12) and 24 (TWA-24) hours post first dose of study medication on Day 1. Positive TWA values represent a reduction in pain intensity
Time Frame: Baseline, 8, 12, and 24 hours post first dose
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale
  Baseline | 3.03 (0.67) | 2.73 (0.62) | 2.84 (0.69) | 2.83 (0.76)
  Change at 8 HR | 0.44 (0.66) | 0.42 (0.55) | 0.59 (0.74) | 0.69 (0.75)
  Change at 12 HR | 0.52 (0.73) | 0.50 (0.58) | 0.71 (0.82) | 0.81 (0.79)
  Change at 24 HR | 0.67 (0.81) | 0.68 (0.66) | 0.89 (0.93) | 0.99 (0.82)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; 8 hour postdose analysis. The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular) and treatment group as factors, and the Patient's Assessment of Pain Intensity at Baseline as a covariate; Test type: Superiority or Other; ANCOVA; Median Difference (Final Values) = 0.09, 95% CI 2-sided [-0.09 to 0.27], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; 8 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.04 to 0.40], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; 8 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.50 to -0.14], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; 8 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.41 to -0.05], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; 8 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.28 to 0.08], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; 12 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.10 to 0.29], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; 12 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.06 to 0.45], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; 12 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.55 to -0.16], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; 12 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.45 to -0.07], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; 12 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.29 to 0.09], Standard Error of Mean 0.10
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; 24 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.08 to 0.35], Standard Error of Mean 0.11
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; 24 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.08 to 0.51], Standard Error of Mean 0.11
Statistical Analysis 13: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; 24 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.61 to -0.18], Standard Error of Mean 0.11
Statistical Analysis 14: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; 24 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.47 to -0.05], Standard Error of Mean 0.11
Statistical Analysis 15: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; 24 hour postdose analysis; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.32 to 0.11], Standard Error of Mean 0.11

9. Secondary Outcome: Number of Participants With ≥30% and ≥50% Reduction From Baseline to Day 2 in Patient's Assessment of Pain Intensity
Description: The Patient's assessment of pain was assessed by completion of the following 5 point scale: My pain over the past 24 hours has been: None (0), Mild (1), Moderate, (2), Severe (3), and Extreme (4).
Time Frame: Baseline, Day 2
Population: ITT and LOCF
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants
  Reduction in Pain Intensity >= 30% | 58 | 69 | 75 | 82
  Reduction in Pain Intensity >= 50% | 43 | 57 | 63 | 71
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; >=30% reduction analyses. The analysis was conducted using analysis of covariance (ANCOVA) with randomization stratum (2 levels: monoarticular or oligoarticular) and treatment group as factors, and the Patient's Assessment of Pain Intensity at Baseline as a covariate; Test type: Superiority or Other; p = 0.0459, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; >=30% reduction analyses; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; >=30% reduction analyses; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; >=30% reduction analyses; Test type: Superiority or Other; p = 0.0410, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; >=30% reduction analyses; Test type: Superiority or Other; p = 0.5592, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; >=50% reduction analyses; Test type: Superiority or Other; p = 0.0277, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; >=50% reduction analyses; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; >=50% reduction analyses; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; >=50% reduction analyses; Test type: Superiority or Other; p = 0.0394, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; >=50% reduction analyses; Test type: Superiority or Other; p = 0.4603, Cochran-Mantel-Haenszel

10. Secondary Outcome: Participant's Assessment of Pain Intensity for the Average Pain Intensity at Baseline
Description: The participant's assessment of pain was assessed by completion of the following 5 point scale: My pain has been: None (0), Mild (1), Moderate, (2), Severe (3), and Extreme (4).
Time Frame: Baseline
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Units on a scale | 3.03 (0.67) | 2.73 (0.62) | 2.84 (0.69) | 2.83 (0.76)

11. Secondary Outcome: Percentage Change From Baseline in the Patient's Assessment of Pain Intensity for the Average Pain Intensity on Days 2-4, Days 2-8 and Days 2-13
Description: The participant's assessment of pain was assessed by completion of the following 5 point scale: My change in pain has been: None (0), Mild (1), Moderate, (2), Severe (3), and Extreme (4). Average change over days was calculated by taking the change from Baseline to the average Pain Intensity score over the days for each patient.
Time Frame: Baseline to Day 13
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Percentage change
  Average change over days 2 - 4 | -44.13 (36.66) | -53.15 (34.17) | -60.11 (33.57) | 2.83 (0.76)
  Average change over days 2 - 8 | -51.36 (35.57) | -61.83 (34.68) | -69.41 (30.86) | -70.05 (27.45)
  Average change over days 2 - 13 | -56.11 (36.47) | -66.26 (35.55) | -73.59 (29.74) | -72.35 (27.39)

12. Secondary Outcome: Number of Participants With Withdrawal From Treatment Due to Lack of Efficacy
Description: Withdrawal due to lack of efficacy was assessed from Days 1 to 8
Time Frame: Day 1 to Day 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants
  Day 1 | 2 | 1 | 0 | 0
  Any time during treatment | 10 | 8 | 4 | 3
  Any time during study | 11 | 9 | 5 | 4
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Withdrawal on Day 1. Pairwise p-values are presented, calculated using Cochran-Mantel-Haenszel statistics, stratified by number of affected joints [1 or >1]) and region; Test type: Superiority or Other; p = 0.5528, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.1779, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.1754, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.3384, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Withdrawal on any time during treatment. Pairwise p-values are presented, calculated using Cochran-Mantel-Haenszel statistics, stratified by number of affected joints [1 or >1]) and region; Test type: Superiority or Other; p = 0.5005, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.0845, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.0213, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.1231, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.6636, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; Withdrawal on any time during study. Pairwise p-values are presented, calculated using Cochran-Mantel-Haenszel statistics, stratified by number of affected joints [1 or >1]) and region; Test type: Superiority or Other; p = 0.5378, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.0818, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.0317, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.1592, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.7956, Cochran-Mantel-Haenszel

13. Secondary Outcome: Participants Global Evaluation of Study Medication Score
Description: The participant rated the study medication that they received during the study by completing the following question:
  How would you rate the study medication you received for pain? 4=Excellent, 3=Good, 2=Fair, 1=Poor
Time Frame: Day 9
Population: ITT
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Scores on a scale | 3.04 (0.87) | 3.11 (0.85) | 3.27 (0.69) | 3.33 (0.75)
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.17 to 0.31], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Celecoxib 800/400 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.02 to 0.46], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.50 to -0.02], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.43 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Celecoxib 800/400 mg vs Indomethacin 50 mg; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.28 to 0.19], Standard Error of Mean 0.12

14. Secondary Outcome: Number of Participants With Pre-specified Gastrointestinal (GI) Adverse Events
Description: The gastrointestinal tolerability was measured by incidence of moderate or severe GI adverse events (nausea, abdominal pain and dyspepsia)
Time Frame: Baseline to Day 14/Early Termination
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants | 1 | 0 | 2 | 3
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; p-value calculated using Cochran-Mantel-Haenszel statistics, stratified by number of affected joints [1; >1], and region; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel

15. Secondary Outcome: Number of Participants With Moderate or Severe Central Nervous System (CNS) Adverse Events
Description: The pre-specfied CNS AEs were headache, nausea, dizziness, vertigo, vomiting and somnolence.
Time Frame: Baseline to Day 14/Early Termination
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Number analyzed (Participants) | 100 | 99 | 96 | 102
Participants | 3 | 2 | 1 | 5
Statistical Analysis 1: Comparison: Celecoxib 50 mg vs Celecoxib 400/200 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.4724, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib 50 mg vs Indomethacin 50 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.7316, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib 400/200 mg vs Indomethacin 50 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.7316, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib 50 mg | Celecoxib 400/200 mg | Celecoxib 800/400 mg | Indomethacin 50 mg
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 0/98 | 1/102
Other Adverse Events (participants affected / at risk) | 22/101 | 22/99 | 21/98 | 32/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 50 mg (N=101) | Celecoxib 400/200 mg (N=99) | Celecoxib 800/400 mg (N=98) | Indomethacin 50 mg (N=102)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 50 mg (N=101) | Celecoxib 400/200 mg (N=99) | Celecoxib 800/400 mg (N=98) | Indomethacin 50 mg (N=102)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 1 | 2 | 1 | 0
Pyrexia (General disorders) | 4 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 4 | 7 | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 6
Headache (Nervous system disorders) | 5 | 4 | 3 | 4
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
Patients Global Evaluation of study medication data was collected at Day 9 only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.